CLINICAL TRIAL: NCT06632405
Title: Camrelizumab Plus Nab-paclitaxel and Anti-histamine Drug Levocetirizine in Metastatic or Recurrent Triple-negative Breast Cancer: a Randomized, Double-arm, Phase 2 Randomized Controlled Trial
Brief Title: A Trial of Camrelizumab Plus Nab-paclitaxel and Levocetirizine in Metastatic or Recurrent TNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Associate Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAnTiH
Record Dates: First submitted 2024-08-27; First posted 2024-10-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; Taxes; levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Camrelizumab+Nab-Paclitaxel+Levocetirizine (Experimental): Camrelizumab 200mg(3mg/kg for patient whose weight is below 50kg) iv, d1, q3w, plus Nab-Paclitaxel 100mg/m2, iv, d1,8,15 q4w, and Levocetirizine 5mg, po, 3 days before 1st administration
  Interventions: Drug: Camrelizumab; Drug: Nab paclitaxel; Drug: Levocetirizine Hydrochloride
- Camrelizumab+Nab-Paclitaxel (Sham Comparator): Camrelizumab 200mg(3mg/kg for patient whose weight is below 50kg) iv, d1, q3w, plus Nab-Paclitaxel 100mg/m2, iv, d1,8,15 q4w
  Interventions: Drug: Camrelizumab; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg (3mg/kg for patient whose weight is below 50kg) will be administered as an intravenous infusion over 30 minutes every three weeks until unacceptable toxic effects or disease progression or other termination criteria appeared.
Drug: Nab paclitaxel — Nab paclitaxel 100mg/m2 will be administered as an intravenous infusion every 4 weeks in d1,8,15until unacceptable toxic effects or disease progression or other termination criteria appeared.
Drug: Levocetirizine Hydrochloride — 5mg daily, start 3 days before the 1st administration
  Arms: Camrelizumab+Nab-Paclitaxel+Levocetirizine

SUMMARY:
This is a phase II, explorative, open-labeled, multi-centered, double-arm, investigator-initiated clinical trial of Camrelizumab (an anti-PD-1 antibody) in combination with Nab-paclitaxel (a chemotherapeutic agent against breast cancer) and Levocetirizine (an antihistamine) in patients with advanced triple-negative breast cancer. 60 subjects will be enrolled in multiple centers. This study aims to evaluate the effects of Camrelizumab combined with Nab-paclitaxel and Levocetirizine in the treatment of advanced TNBC.

DETAILED DESCRIPTION:
This is a phase II, explorative, open-labeled, multi-centered, double-arm, investigator-initiated clinical trial to evaluate the effects of Camrelizumab combined with Nab-paclitaxel and Levocetirizine in the treatment of advanced TNBC. The study aims to enroll 60 subjects in multiple centers. The primary objective is to assess the overall response rate (ORR). All enrolled patients will be treated with Camrelizumab 200mg (iv. 3mg/kg for patient whose weight is below 50kg) on day 1 of each 3 week, and Nab-paclitaxel 100mg/m2, iv, on d1,8,15 of each 4 week, in combination with Levocetirizine of 5mg, po., 3 days before 1st administration.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the written informed consent;
2. Aged ≥ 18 and ≤ 70 years old;
3. Confirmed recurrent and metastatic triple negative breast cancer by imaging and pathology (ER negative (IHC ER positive percentage < 1%), PR negative (IHC PR positive percentage < 1%), HER2 negative (IHC -/+or IHC++but FISH/CISH -)), at least one measurable focus meeting the RECIST v1.1 standard;
4. Untreated local recurrence of unresectable TNBC or untreated distant metastasis of TNBC
5. Must be able to swallow tablets;
6. Clarify the positive status of PD-L1 expression and CPS score ≥ 1
7. ECOG score: 0 to 1;
8. Expected survival period ≥ 12 weeks;
9. The results of patient's blood tests are as follows (excluding the use of any blood components and cell growth factors during screening):

   * Absolute neutrophil count ≥ 1.5 × 109/L;
   * Platelets ≥ 100 × 109/L;
   * Hemoglobin ≥ 9g/dL;
   * Serum albumin ≥ 3g/dL;
   * Thyroid stimulating hormone (TSH) ≤ ULN (if abnormal, T3 and T4 levels should be examined simultaneously. If T3 and T4 levels are normal, they can be included in the group);
   * Bilirubin ≤ 1.0 times ULN (Gilbert's syndrome or liver metastasis subject total bilirubin ≤ 1.5 times ULN);
   * ALT and AST ≤ 1.5 times ULN (liver metastasis subjects ≤ 3 times ULN);
   * AKP ≤ 2.5 times ULN;
   * Renal function within 7 days before the first administration: serum creatinine ≤ 1.5 times ULN or creatinine clearance rate ≥ 60mL/min (using the standard Cockcroft Gault formula, see Appendix 3);
10. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 6 months after the last dose of study treatment.
11. Left ventricular ejection fraction ≥ 50%

Exclusion Criteria:

1. Received other interventional clinical trials within 28 days before the first dose;
2. Failure to recover from adverse reactions of previous treatment
3. Neurological disorders of grade ≥ 2
4. Untreated active brain metastases or meningeal metastases
5. Previously received nab-paclitaxel neoadjuvant therapy or adjuvant therapy and experienced local recurrence or distant metastasis within 12 months;
6. Has experienced severe allergic reactions to other monoclonal antibodies;
7. Received other anti-tumor treatments within 28 days before the first administration;
8. Suffering from hypertension and unable to achieve good control with antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
9. Received antibody or T cell co stimulatory therapy such as PD-1, PD-L1, PD-L2, CTLA-4, Tim3, LAG3, etc;
10. Special genetic diseases (including rare galactose intolerance, primary lactase deficiency, or glucose galactose malabsorption);
11. Active autoimmune disease or history of autoimmune disease (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or complete remission of childhood asthma without any intervention in adulthood may be included; subjects with asthma requiring medical intervention with bronchodilators may not be included);
12. Heart diseases, such as:

    * NYHA grade 2 or above heart failure
    * Unstable angina pectoris
    * Have experienced a myocardial infarction within the past year
    * Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention；
13. Urine protein level is ≥++, or the 24-hour urine protein level is ≥ 1.0 g;
14. Known genetic or acquired bleeding and thrombophilia tendencies (such as hemophilia patients, coagulation dysfunction, thrombocytopenia, splenomegaly, etc.);
15. Have a history of tuberculosis;
16. Active period of HBV or HCV, and other active infectious diseases;
17. Had or is currently experiencing qualitative pneumonia or requires steroid treatment for pneumonia;
18. Congenital or acquired immune dysfunction (such as HIV infected individuals);
19. Received or about to receive a live vaccine within 4 weeks prior to the study or possibly during the study period;
20. Allergic or contraindicated to the experimental drug.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | from the first drug administration up to the first occurrence of progression or death （up to 36 weeks）
  The propotion of subjects with CR or PR.

SECONDARY OUTCOMES:
Adverse events/Serious adverse events | from the first drug administration to within 90 days for the last dose
  Adverse events/Serious adverse events
Disease Control Rate (DCR) | from the first drug administration up to the first occurrence of progression or death （up to 36 weeks）
  The propotion of subjects with CR, PR, or SD.
Clinical benefit rate (CBR) | propotion of subjects with CR, PR, or SD for >=6 months （up to 36 weeks）
  The propotion of subjects with CR, PR, or SD for >=6 months during the study
Duration of response (DoR) | from the first drug administration up to the first occurrence of progression or death （up to 36 weeks）
  The time from randomization to disease progression or death for patients who achieve complete or partial alleviation
Time to response (TTR) | from the first drug administration up to the first occurrence of progression （up to 36 weeks）
  Time from date of first dose to date of first occurrence of response
Progression-Free-Survival (PFS) | from the first drug administration up to the first occurrence of progression or death （up to 36 weeks）
  from the first drug administration up to the first occurrence of progression or death (up to 24 months)
Overall survival (OS) | 12 months after the first drug administration
  12 months after the first drug administration
Biomarkers | pre-treatment, up to 24 months
  Compare the change of biomarkers from urine, blood or tissues, such as the carcinoembryonic antigen (ug/L), before or after the treatments.
Biomarkers | pre-treatment, up to 24 months
  Compare the change of biomarkers from urine, blood or tissues, such as the CA125/199/153(u/ml), before or after the treatments.
patient reported outcomes (PRO) | during the study and up to 36 weeks after the end
  direct reports from patients about their health, the scale Quality of Life questionnaire (QLQ)-BR23/C30 will be used for assecessment. Higher score indicate better life quality

CONTACTS AND LOCATIONS:
Overall Officials: Jieqiong Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University